CLINICAL TRIAL: NCT05837923
Title: Radicle™ Relief 2: A Randomized, Blinded, Placebo-Controlled Direct-to-Consumer Study of Health and Wellness Products on Pain and Other Health Outcomes
Brief Title: Radicle Relief 2: A Study of Health and Wellness Products on Pain and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-2303
Record Dates: First submitted 2023-04-06; First posted 2023-05-01 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2024-11

CONDITIONS: Pain; Neuropathic Pain; Nociceptive Pain
MeSH Terms: conditions — Pain; Neuralgia; Nociceptive Pain

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' study product assignment. Participants are blinded to the study product they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Placebo Control 1 (Placebo Comparator): Relief Product Form 1 - control
  Interventions: Dietary Supplement: Placebo Control Form 1
- Active Product 1.1 (Experimental): Relief Product Form 1 - active product 1
  Interventions: Dietary Supplement: Relief Active Study Product 1.1 Usage
- Active Product 1.2 (Experimental): Relief Product Form 1 - active product 2
  Interventions: Dietary Supplement: Relief Active Study Product 1.2 Usage
- Placebo Control 2 (Placebo Comparator): Relief Product Form 2 - control
  Interventions: Dietary Supplement: Placebo Control Form 2
- Active Product 2.1 (Experimental): Relief Product Form 2 - active product 1
  Interventions: Dietary Supplement: Relief Active Study Product 2.1 Usage
- Placebo Control 3 (Placebo Comparator): Relief Product Form 3 - control
  Interventions: Dietary Supplement: Placebo Control Form 3
- Active Product 3.1 (Experimental): Relief Product Form 3 - active product 1
  Interventions: Dietary Supplement: Relief Active Study Product 3.1 Usage
- Active Product 3.2 (Experimental): Relief Product Form 3 - active product 2
  Interventions: Dietary Supplement: Relief Active Study Product 3.2 Usage
- Active Product 3.3 (Experimental): Relief Product Form 3 - active product 3
  Interventions: Dietary Supplement: Relief Active Study Product 3.3 Usage

INTERVENTIONS:
Dietary Supplement: Relief Active Study Product 1.1 Usage — Participants will use their Radicle Relief Active Study Product 1.1 as directed for a period of 6 weeks.
  Arms: Active Product 1.1
Dietary Supplement: Relief Active Study Product 1.2 Usage — Participants will use their Radicle Relief Active Study Product 1.2 as directed for a period of 6 weeks.
  Arms: Active Product 1.2
Dietary Supplement: Placebo Control Form 1 — Participants will use their Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo Control 1
Dietary Supplement: Relief Active Study Product 2.1 Usage — Participants will use their Radicle Relief Active Study Product 2.1 as directed for a period of 6 weeks.
  Arms: Active Product 2.1
Dietary Supplement: Placebo Control Form 2 — Participants will use their Placebo Control Form 2 as directed for a period of 6 weeks.
  Arms: Placebo Control 2
Dietary Supplement: Placebo Control Form 3 — Participants will use their Placebo Control Form 3 as directed for a period of 6 weeks.
  Arms: Placebo Control 3
Dietary Supplement: Relief Active Study Product 3.1 Usage — Participants will use their Radicle Relief Active Study Product 3.1 as directed for a period of 6 weeks.
  Arms: Active Product 3.1
Dietary Supplement: Relief Active Study Product 3.2 Usage — Participants will use their Radicle Relief Active Study Product 3.2 as directed for a period of 6 weeks.
  Arms: Active Product 3.2
Dietary Supplement: Relief Active Study Product 3.3 Usage — Participants will use their Radicle Relief Active Study Product 3.3 as directed for a period of 6 weeks.
  Arms: Active Product 3.3

SUMMARY:
A randomized, blinded, placebo-controlled study assessing the impact of health and wellness products on pain and other health outcomes

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled study conducted with adult participants, age 21 and older and residing in the United States.

Eligible participants will (1) endorse a desire for less pain, (2) indicate an interest in taking a health and wellness product to potentially help their pain, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants with known liver or kidney disease, heavy drinkers, and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Those taking certain medications will be excluded.

Self-reported data are collected electronically from eligible participants over 7 weeks. Participant reports of health indicators will be collected during baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21 years of age and older at the time of electronic consent, inclusive of all ethnicities, races, genders and/or gender identities
* Resides in the United States
* Endorses less pain as a primary desire
* Selects pain and/or looking to improve their pain as a reason for their interest in taking a health and wellness product
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Reports being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* The calculated validated health survey (PRO) score during enrollment represents less than mild severity
* Reports a diagnosis of liver or kidney disease
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports current enrollment in a clinical trial
* Lack of reliable daily access to the internet
* Reports current or recent (within 3 months) use of chemotherapy or immunotherapy
* Reports taking medications with a known moderate or severe interaction with any of the active ingredients studied, or a substantial safety risk: Anticoagulants, a medication that warns against grapefruit consumption, corticosteroids at doses greater than 5 mgs per day, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, or MAOIs (monoamine oxidase inhibitors)
* Reports a diagnosis of heart disease when a known contraindication exists for any of the active ingredients studied: NYHA (New York Heart Association) Class III or IV congestive heart failure, Atrial fibrillation, Uncontrolled arrhythmias

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2016 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Change in pain interference | 6 weeks
  Mean difference in pain interference score as assessed by Patient Reported Outcome Measurement System (PROMIS) Pain Interference 6A (scale 6-30; with higher scores corresponding to greater pain interference)

SECONDARY OUTCOMES:
Change in neuropathic pain | 6 weeks
  Mean difference in neuropathic pain score as assessed by PROMIS Neuropathic Pain 5A (scale 5-25; with higher scores corresponding to greater neuropathic pain)
Change in nociceptive pain | 6 weeks
  Mean difference in nociceptive pain score as assessed by PROMIS Nociceptive Pain 5A (scale 5-25; with higher scores corresponding to greater nociceptive pain)
Change in pain intensity | 6 weeks
  Mean difference in pain intensity score as assessed by PROMIS Pain Intensity 1A (scale 1-10; with 0 being 'No pain' and 10 being 'The worst imaginable pain')
Change in feelings of anxiety | 6 weeks
  Mean difference in anxiety score as assessed by PROMIS Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Change in sleep | 6 weeks
  Mean difference in sleep score as assessed by PROMIS Sleep Disturbance Form 4A (scale 4-20; with higher scores corresponding to more severe sleep disturbance)
Change in energy (fatigue) | 6 weeks
  Mean difference in fatigue score as assessed by PROMIS Fatigue 4A (scale 4-20; with higher scores corresponding to greater fatigue)
Minimal clinically important difference (MCID) in pain interference | 6 weeks
  Likelihood of experiencing MCID in pain interference score as assessed by PROMIS Pain Interference 6A
Minimal clinically important difference (MCID) in neuropathic pain | 6 weeks
  Likelihood of experiencing MCID in neuropathic pain score as assessed by PROMIS Neuropathic Pain 5A
Minimal clinically important difference (MCID) in nociceptive pain | 6 weeks
  Likelihood of experiencing MCID in nociceptive pain score as assessed by PROMIS Nociceptive Pain 5A
Minimal clinically important difference (MCID) in pain intensity | 6 weeks
  Likelihood of experiencing MCID in pain intensity score as assessed by PROMIS Pain Intensity 1A

OTHER OUTCOMES:
Change in focus (cognitive function) | 6 weeks
  Mean difference in cognitive function score as assessed by PROMIS Cognitive Function 4A (scale 4-20; with higher scores corresponding to greater cognitive function)
Change in mood (emotional distress-depression) | 6 weeks
  Mean difference in emotional distress score as assessed by PROMIS Emotional Distress- Depression 4A (scale 4-20; with higher scores corresponding to greater levels of emotional distress)
Change in libido | 6 weeks
  Mean difference in libido score as assessed by PROMIS Sexual Interest 2.0 (scale 2-10; with higher scores corresponding to greater interest in sexual activity)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com